CLINICAL TRIAL: NCT00001668
Title: Endolymphatic Sac Tumors in a Population of Patients With Von Hippel-Lindau Disease:The Natural History and Pathobiology, and a Prospective Non-Randomized Clinical Trial of Hearing Preservation Surgery in Patients With Early Stage Endolymphatic Sac Tumors
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970102; 97-N-0102
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Deafness; Kidney Diseases; Kidney Neoplasms; Neoplasms; Retinal Diseases
Keywords: Deafness; Hemangioblastoma; Papillary Carcinoma; VHL Gene; Vestibular Function; von Hippel-Lindau Disease
MeSH Terms: conditions — Deafness; Kidney Diseases; Kidney Neoplasms; Neoplasms; Retinal Diseases; Hemangioblastoma; Carcinoma, Papillary; von Hippel-Lindau Disease

SUMMARY:
The von Hippel Lindau (VHL) gene has recently been identified as the genetic defect resulting in a syndrome of multiple neoplasias. Patients with VHL disease develop retinal angiomata, renal cysts and/or carcinomas, CNS hemangioblastomas as well as pancreatic cysts and pheochromocytomas. Investigators have shown the gene to be a tumor suppressor type proto-oncogene located at chromosomal locus 3p26. The gene includes three exons whose gene product targets a cellular transcription factor Elongin SIII. Binding of the VHL proteins to two subunits of this elongation factor inhibits transcription and may play a crucial role in the clinical development of the von Hippel Lindau phenotype.

DETAILED DESCRIPTION:
The von Hippel Lindau (VHL) gene has recently been identified as the genetic defect resulting in a syndrome of multiple neoplasias. Patients with VHL disease develop retinal angiomata, renal cysts and/or carcinomas, CNS hemangioblastomas as well as pancreatic cysts and pheochromocytomas. Investigators have shown the gene to be a tumor suppressor type proto-oncogene located at chromosomal locus 3p26. The gene includes three exons whose gene product targets a cellular transcription factor Elongin SIII. Binding of the VHL proteins to two subunits of this elongation factor inhibits transcription and may play a crucial role in the clinical development of the von Hippel Lindau phenotype.

ELIGIBILITY:
Patients meeting the diagnostic criteria for von Hippel-Lindau (VHL) disease.

No persons who are pregnant or lactating are eligible for the surgical arm of this protocol until the pregnancy and/or nursing period has reached completion.

No patients with disorders associated with multiple abnormalities of the middle ear and inner ear. Specific laboratory abnormalities such as anti-HIV-1, FTA-Abs, serum ANA, and ANCA have been associated with AIDS, Syphilis, Systemic Lupus Erythematosus, and Wegener's Granulomatosis, respectively.

No patients currently undergoing chemotherapeutic regimen with ototoxic agents (e.g., cisplatin). Other agents will be reviewed on a case-by-case basis for their potential to cause ototoxicity and thereby interfere with audiologic data interpretation.

Patients with an ELST in an only hearing ear will be excluded from the protocol for surgical treatment of ELST's (except in cases where other medical indications necessitate intervention for the welfare of the patient).

Patients with only unilateral vestibular function on the side affected by the ELST, as documented by caloric ENG testing, will be excluded from the surgical treatment group in most cases.

No patients with the inability to understand all of the requirements of the study or inability to give informed consent and/or comply with all aspects of the evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1997-04; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States